CLINICAL TRIAL: NCT04684342
Title: Predictors of Fungal Infection in Non-neutropenic Patients in Intensive Care Units
Brief Title: Fungal Infection in Patients in Intensive Care Units
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdou Mahmoud, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Fungal infection in ICU
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cirrhotic ICU Patients (Experimental): about 150 patients with cirrhosis fulfill- ing the inclusion criteria that will be admitted to Tropical Medicine and Gas- troenterology Department, Al-Rajhi Liver Hospital, Assiut University Hospi- tals) will be evaluated for fungal infection.
  Interventions: Diagnostic Test: Routine Laboratory investigations

INTERVENTIONS:
Diagnostic Test: Routine Laboratory investigations — 1. Complete blood picture
  2. Liver function test and prothrombine time & concentration.
  3. Blood urea and creatinine
  4. Blood glucose, serum Na and K
  5. CRP and ESR
  6. Clinical specimens will be collected from patients according to the suspected site of infection (e.g. blood, urine, ascitic fluid, sputum or endo- tracheal aspirates) VITEK 2Compact inflammatory markers

SUMMARY:
Predictors of fungal infection in non-neutropenic patients in intensive care units and the aim of the study is To evaluate the frequency of fungal infection in non-neutropenic patients in Intensive Care Units.

To evaluate the risk factors of fungal infection in these patients.

DETAILED DESCRIPTION:
The incidence of candidemia in the overall population ranges from 1.7 to 10 episodes per 100,000 inhabitants and Candida is one of the ten leading causes of bloodstream infections in developed countries. An estimated 33-55% of all episodes of candidemia occur in intensive care units (ICU) and are associated with mortality rates ranging from 5% to 71%. Candida fungemia may have an endogenous or an exogenous origin, and in recent years a growing proportion of episodes of candidemia have been caused by Candida species other than albicans. The most important independent conditions predisposing to candidemia in ICU patients include prior abdominal surgery, intravascular catheters, acute renal failure, parenteral nutrition, broad-spectrum antibiotics, a prolonged ICU stay, the use of corticosteroids and mucosal colonization with Candida. In recent years, several studies have shown that ICU patients with mucosal Candida colonization, particularly if multifocal, are at a higher risk for invasive candidiasis, and that colonization selects a population amenable to antifungal prophylaxis or empirical therapy. Candidemia in ICUs is associated with a con- siderable increase in hospital costs and length of hospital stay.

Invasive fungal infection (IFI) is a grave infection associated with serious effects in patients with chronic diseases including liver cirrhosis. The diagnosis of IFI re- quires histopathological evidence of tissue invasion, or isolation in blood cultures, or isolation from a normally sterile body fluid or site, with samples collected intra-op- eratively or by percutaneous needle aspiration. Awareness of IFI has been increased in clinical practice with the increased survival of patients in immunocompromised states. Such infections are associated with a high morbidity and significant mortality, requiring early diagnosis and appropriate treatment, but also optimal prophylaxis in patients at high risk.

Globally, several studies had assessed fungal infections in non-neutropenic patients, however, to our knowledge, searching for fungal infections in these patients are un- derestimated in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with liver cirrhosis that will be clinically suspected to have in- fection.

Exclusion Criteria:

* Age < 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
frequency of fungal infection in cirrhotic patients | 4 months
  frequency of fungal infection in cirrhotic patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zakaria, Professor, Study Chair — Assiut University

REFERENCES:
- [Background] Leon DA, McCambridge J. Liver cirrhosis mortality rates in Britain from 1950 to 2002: an analysis of routine data. Lancet. 2006 Jan 7;367(9504):52-6. doi: 10.1016/S0140-6736(06)67924-5. PMID 16399153
- [Background] Runyon BA; AASLD. Introduction to the revised American Association for the Study of Liver Diseases Practice Guideline management of adult patients with ascites due to cirrhosis 2012. Hepatology. 2013 Apr;57(4):1651-3. doi: 10.1002/hep.26359. No abstract available. PMID 23463403
- [Background] Bucsics T, Schwabl P, Mandorfer M, Peck-Radosavljevic M. Prognosis of cirrhotic patients with fungiascites and spontaneous fungal peritonitis (SFP). J Hepatol. 2016 Jun;64(6):1452-4. doi: 10.1016/j.jhep.2016.01.039. Epub 2016 Feb 23. No abstract available. PMID 26916528